CLINICAL TRIAL: NCT00700271
Title: Efficacy of a Combination of Amlodipine / Valsartan on Blood Pressure Control, With One Nocturnal or Diurnal Intake a Day, in Ambulatory Blood Pressure Monitoring Setting, in Essential Uncontrolled Hypertensive Patients With Amlodipine 5mg ; The ExPERT Study
Brief Title: Efficacy of a Combination of Amlodipine/Valsartan on 24H Blood Pressure Control With One Nocturnal or Diurnal Intake a Day
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CVAA489AFR01
Record Dates: First submitted 2007-12-11; First posted 2008-06-18 (Estimated); Results first posted 2011-01-06 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2011-05

CONDITIONS: Hypertension
Keywords: Hypertension; ambulatory blood pressure monitoring
MeSH Terms: conditions — Hypertension | interventions — Amlodipine; Valsartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Morning Intake (Experimental): After randomization, participants received a single daily oral dose of 5 mg amlodipine and 160 mg valsartan free combination therapy, taken in the morning between 6-10 am. At week 4, uncontrolled patients (msSBP >= 140 mmHg and/or msDBP >= 90 mmHg or msSBP >= 130 mmHg and/or msDBP >= 80 mmHg in the case of diabetes or renal insufficiency measured by using conventional methods) received amlodipine/valsartan 10/160 mg for 4 additional weeks. Patients who were controlled at Week 4 (msSBP < 140 mmHg and msDBP < 90 mmHg or msSBP < 130 mmHg and msDBP < 80 mmHg in the case of diabetes or renal insufficiency) continued their amlodipine/valsartan 5/160 mg treatment for the remaining 4 weeks of the study.
  Interventions: Drug: Amlodipine; Drug: Valsartan
- Evening Intake (Experimental): After randomization participants received a single daily oral dose of 5 mg amlodipine and 160 mg valsartan free combination therapy, taken in the evening between 6-10 pm. At week 4, uncontrolled patients (msSBP >= 140 mmHg and/or msDBP >= 90 mmHg or msSBP >= 130 mmHg and/or msDBP >= 80 mmHg in the case of diabetes or renal insufficiency measured by using conventional methods) received amlodipine/valsartan 10/160 mg for 4 additional weeks. Patients who were controlled at Week 4 (msSBP < 140 mmHg and msDBP < 90 mmHg or msSBP < 130 mmHg and msDBP < 80 mmHg in the case of diabetes or renal insufficiency) continued their amlodipine/valsartan 5/160 mg treatment for the remaining 4 weeks of the study.
  Interventions: Drug: Amlodipine; Drug: Valsartan

INTERVENTIONS:
Drug: Amlodipine — 5 mg or 10 mg tablets.
Drug: Valsartan — 160 mg capsules.

SUMMARY:
This study was a multicenter, randomized, PROBE-type (prospective, randomized, open label, blinded end-point) study of 12 weeks duration comprising four visits, carried out in patients with essential arterial hypertension not controlled on four weeks treatment with amlodipine 5 mg alone.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Essential uncontrolled or naive hypertensive patients (SBP ≥= 140 mmHG, DBP - >/=90 mm Hg, or SBP >= 130 mmHg, DBP >= 80 mmHg if diabetes or renal impairment) except patients treated with amlodipine, or intolerant of ARBs and/or calcium channel blockers.

Exclusion Criteria:

* Severe hypertension : SBP >= 180 mmHg, DBP >= 110mmHg
* Pregnancy
* Allergia to ARBs and/or to calcium channel blockers
* Antihypertensive tritherapy at V1
* History of heart failure, pectoris angina, stroke, myocardial infarction
* Diabetes type I
* Renal impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 478 (Actual)
Dates: Start 2007-10; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roland Asmar, Principal Investigator — principle investigator; Institut cardiovasculaire 75016 Paris
Locations (2):
- Investigative sites in France, Paris, France
- Investigative sites in Tunisia, Tunisia, Tunisia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eligible patients entered a 4-week open-label amlodipine screening phase with amlodipine 5 mg taken orally once a day. At the end of the screening phase, patients whose blood pressure was not adequately controlled (defined as SBP/DBP >= 125/80 mmHg 24-hr mean) on ambulatory blood pressure monitoring were randomized to one of two treatment groups.
Period: Overall Study
Arm/Group | Morning Intake | Evening Intake
Started | 278 | 268
Completed | 264 | 256
Not Completed | 14 | 12
Not completed — Adverse Event | 4 | 6
Not completed — Protocol Violation | 1 | 0
Not completed — Administrative Reasons | 1 | 0
Not completed — Withdrawal by Subject | 6 | 4
Not completed — Lost to Follow-up | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Morning Intake | Evening Intake | Total
Number analyzed (Participants) | 242 | 237 | 479
Age Continuous [Mean (Standard Deviation); unit: years] — Demographic data is provided for the Intent-to-Treat population, which included all the patients randomized and treated in the study and for whom two ABPM evaluations were available.
  years | 55.8 (9.89) | 56.2 (9.59) | 56.0 (9.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 114 | 111 | 225
  Male | 128 | 126 | 254

OUTCOME MEASURES:

1. Primary Outcome: Absolute Reduction From Baseline in 24-hour Mean Systolic Blood Pressure (SBP) on Ambulatory Blood Pressure Monitoring
Description: Ambulatory Blood Pressure Monitoring (ABPM) over a 30-hour period was carried out in all patients at two visits during the study, 72 hours before visit 2 (baseline) and visit 4 (week 8). ABPM for visit 2 was carried out prior to randomization and the first dose of the amlodipine/valsartan combination study therapy. ABPM for visit four began after 12 weeks of treatment and before the last office blood pressure was taken. Covariates included baseline level, country, up-titration + treatment*country and treatment*up-titration interactions in case statistically significant at a 0.10 level.
Time Frame: Baseline (Week 0, after completion of screening period) and Week 8 (after 8 weeks of combination therapy)
Population: The Intent-to-treat (ITT) population included all patients randomized and treated in the study and for whom two Ambulatory Blood Pressure Monitoring (ABPM) evaluations are available.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Morning Intake | Evening Intake
Number analyzed (Participants) | 242 | 237
mmHg | -12.01 (0.70) | -11.3 (0.71)

2. Secondary Outcome: Absolute Reduction From Baseline in Diurnal Mean Systolic Blood Pressure (SBP)/Diastolic Blood Pressure (DBP) on Ambulatory Blood Pressure Monitoring
Description: as for outcome 1
Time Frame: Baseline (Week 0, after completion of screening period) and Week 8 (after 8 weeks of combination therapy)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Morning Intake | Evening Intake
Number analyzed (Participants) | 242 | 237
mmHg
  Systolic Blood Pressure (SBP) | -13.50 (0.78) | -11.99 (0.8)
  Diastolic Blood Pressure (DBP) | -7.56 (0.49) | -7.11 (0.5)

3. Secondary Outcome: Absolute Reduction From Baseline in Nocturnal Mean Systolic Blood Pressure (SBP)/Diastolic Blood Pressure (DBP) on Ambulatory Blood Pressure Monitoring
Description: as for outcome 1
Time Frame: Baseline (Week 0, after completion of screening period) and Week 8 (after 8 weeks of combination therapy)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Morning Intake | Evening Intake
Number analyzed (Participants) | 242 | 237
mmHg
  Systolic Blood Pressure (SBP) | -9.68 (0.74) | -10.33 (0.76)
  Diastolic Blood Pressure (DBP) | -5.01 (0.46) | -6.3 (0.47)

4. Secondary Outcome: Absolute Reduction From Baseline in 24-hour Mean Diastolic Blood Pressure (DBP) on Ambulatory Blood Pressure Monitoring
Description: as for outcome 1
Time Frame: Baseline (Week 0, after completion of screening period) and Week 8 (after 8 weeks of combination therapy)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Morning Intake | Evening Intake
Number analyzed (Participants) | 242 | 237
mmHg | -6.53 (0.42) | -6.79 (0.43)

5. Secondary Outcome: Absolute Reduction From Baseline in 6-hour Mean Systolic Blood Pressure (SBP)/Diastolic Blood Pressure (DBP) on Ambulatory Blood Pressure Monitoring
Description: as for outcome 1
Time Frame: Baseline (Week 0, after completion of screening period) and Week 8 (after 8 weeks of combination therapy)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Morning Intake | Evening Intake
Number analyzed (Participants) | 242 | 237
mmHg
  Systolic Blood Pressure (SBP) | -12.16 (0.88) | -11.37 (0.90)
  Diastolic Blood Pressure (DBP) | -7.71 (0.59) | -7.01 (0.60)

6. Secondary Outcome: Mean Seated Systolic Blood Pressure (msSBP)/Mean Seated Diastolic Blood Pressure (msDBP) Variation Between Week 0 and Week 8 in Office Blood Pressure
Description: At each of the office visits, blood pressure was recorded in the morning between 08.00 and 11.00, before any antihypertensive treatment was taken. The patient remained in a sitting position for five minutes; the investigator then took three blood pressure and one pulse rate reading. The measurements were recorded at 1-2 minute intervals. Covariates included baseline level, country, up-titration + treatment*country and treatment*up-titration interactions in case statistically significant at a 0.10 level.
Time Frame: Baseline (Week 0, after completion of screening period) and Week 8 (after 8 weeks of combination therapy)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Morning Intake | Evening Intake
Number analyzed (Participants) | 231 | 232
mmHg
  Systolic Blood Pressure (SBP) | -18.7 (0.9) | -17.3 (0.9)
  Diastolic Blood Pressure (DBP) | -10.1 (0.6) | -8.6 (0.7)

7. Secondary Outcome: Mean Seated Systolic Blood Pressure (msSBP)/Mean Seated Diastolic Blood Pressure (msDBP) Variation Between Week -4 to Week 8 in Office Blood Pressure
Description: as for outcome 6
Time Frame: Screening visit (Week -4, prior to 4-week open-label screening phase) and Week 8 (after 8 weeks of combination therapy)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Morning Intake | Evening Intake
Number analyzed (Participants) | 231 | 232
mmHg
  Systolic Blood Pressure (SBP) | -32.2 (1.1) | -29 (1.2)
  Diastolic Blood Pressure (DBP) | -16.6 (0.8) | -14.3 (0.8)

8. Secondary Outcome: Percentage of Participants With 24-hour Mean Systolic Blood Pressure (SBP)/Diastolic Blood Pressure (DBP) < 125/80 mmHg at Endpoint With Ambulatory Blood Pressure Monitoring
Description: Ambulatory Blood Pressure Monitoring (ABPM) over a 30-hour period was carried out in all patients at two visits during the study, 72 hours before visit 2 (baseline) and visit 4 (week 8). ABPM for visit four began after 12 weeks of treatment and before the last office blood pressure was taken.
Time Frame: Visit 4 (week 8)
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Morning Intake | Evening Intake
Number analyzed (Participants) | 242 | 237
Percentage of Participants | 47.6 | 46.9

9. Secondary Outcome: Percentage of Participants With Diurnal Mean Systolic Blood Pressure (SBP)/Diastolic Blood Pressure (DBP) < 135/85 mmHg at Endpoint With Ambulatory Blood Pressure Monitoring
Description: as for outcome 8
Time Frame: Visit 4 (week 8)
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Morning Intake | Evening Intake
Number analyzed (Participants) | 242 | 237
Percentage of Participants | 65.3 | 58.2

10. Secondary Outcome: Percentage of Participants With Nocturnal Mean Systolic Blood Pressure (SBP)/Diastolic Blood Pressure (DBP) < 120/70 mmHg at Endpoint With Ambulatory Blood Pressure Monitoring
Description: as for outcome 8
Time Frame: Visit 4 (week 8)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Morning Intake | Evening Intake
Number analyzed (Participants) | 242 | 237
Percentage of participants | 41.3 | 46.8

11. Secondary Outcome: Percentage of Participants With Controlled Office Mean Seated Systolic Blood Pressure (msSBP)/Mean Seated Diastolic Blood Pressure (msDBP) at Endpoint
Description: At each of the office visits, blood pressure was recorded in the morning between 08.00 and 11.00, before any antihypertensive treatment was taken. The patient remained in a sitting position for 5 minutes; the investigator then took 3 blood pressure and 1 pulse rate reading. The measurements were recorded at 1-2 minute intervals. BP Control is defined as msSBP/msDBP <149/90 mmHg and/or <130/80 mmHg if diabetes or renal insufficiency (RI).
Time Frame: Visit 4 (week 8)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Morning Intake | Evening Intake
Number analyzed (Participants) | 242 | 237
Percentage of participants | 71.1 | 72.6

ADVERSE EVENTS:
Arm/Group | Morning Intake | Evening Intake
Serious Adverse Events (participants affected / at risk) | 2/278 | 2/268
Other Adverse Events (participants affected / at risk) | 0/278 | 0/268
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Morning Intake (N=278) | Evening Intake (N=268)
Atrial fibrillation (Cardiac disorders) | 1 | 0
Atrioventricular block (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Stress (Psychiatric disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial; or publication of the trial results in their entirety.